CLINICAL TRIAL: NCT02450604
Title: Prevalence of Fabry's Disease in a Population of Patients With Chronic Pain
Acronym: DOUFABIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2014/23
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Fabry's Disease; Chronic Pain
Keywords: Prevalence Study; Fabry's disease; Chronic pain
MeSH Terms: conditions — Fabry Disease; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with chronic pains of unknown aetiology (Other)
  Interventions: Genetic: Diagnosis of Fabry disease

INTERVENTIONS:
Genetic: Diagnosis of Fabry disease — The diagnosis of Fabry disease necessitates biochemical enzymatic measures of alphagalactosidase A activity in males, and genetic analysis using direct sequencing of GLA in females.

SUMMARY:
Fabry disease is a rare inherited metabolic disorder that predominantly affects heart, kidneys and nervous system. Fabry disease has been searched in series of patients presenting different isolated signs caused by the affection of one of these organs. Acroparesthesias and chronic crises of pain of different origins are reported in the large majority of patients during the progression of the disease. Moreover, this signs are frequently inaugurating the disease. The investigators have previously performed a preliminary single-center study which permitted to identify one female patient with Fabry disease in a series of 147 consecutive patients with chronic pain tested. The investigators now propose to confirm the results of our preliminary study. The investigators plan to evaluate the prevalence of Fabry disease in a series of 1000 patients suffering from chronic pains of undetermined aetiology and consecutively recruited.

DETAILED DESCRIPTION:
Fabry disease (FD) is a rare X-linked multisytemic lysosomal disorder caused by alpha-galactosidase deficiency. Globotriaosylcéramide (Gb3) deposits are observed in almost all tissues examined. Signs of the disease appear earlier and are more severe in affected males than in females. Myocardiopathy, renal failure and neurological signs including chronic pain and peripheral neuropathies are the most frequent signs. The availability of two enzymatic replacement therapies now provides a specific and effective treatment for patients. The prevalence of FD is estimated between 1/40,000 and 1/117,000. The frequency of Fabry disease has previously been estimated in several series of patients presenting one single sign, ie renal failure, hypertrophic myocardiopathy and early onset stroke. However, no data are available about the prevalence of FD in populations of patients suffering from chronic pains of unknown origin.

The diagnosis of FD will be performed by standard procedures following international recommendations. These require the search for a deficiency of alphagalactosidase A activity on leucocytes in males and genetic analysis of the GLA gene in females (Germain et al. 2010).

The patients in whom the diagnosis of FD is established during this study, will be call in for an additional visit in the Investigating Centre in order to confirm the diagnosis and propose suitable assessment and care.

ELIGIBILITY:
Inclusion Criteria:

* patients of both sex,
* aged from 6 to 80,
* with chronic pains of unknown aetiology including: acroparesthesias, and/or pain crises evolving more than 3 months, continued neuropathic evolving more than 3 months, and/or multiple pains evolving more than 3 months and/or recurrent abdominal crises of pain who come for a clinical visit in the pain Centres of France.

Exclusion Criteria:

* chronic pain of known cause

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Fabry disease in one patient suffering from chronic pains | J1 to 2 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Cyril GOIZET, Principal Investigator — University Hospital, Bordeaux
Locations (21):
- France (21):
  - Cs douleur chronique GHSR, CHU Sud Réunion, Saint-Pierre, La Réunion
  - CeRCa, Unité de Neuromyologie, CHU de Fort de France, FORT de France, Martinique
  - Centre Douleurs Chroniques, CH de la Côte Basque, Bayonne
  - Centre Douleurs Chroniques, CHU de Bordeaux, Bordeaux
  - Service de médecine Polyvalent, CH de La Dracénie, Draguignan
  - Anesthésie, Hôpital Raymond Poincaré, Garches
  - Centre de la douleur de l'Adulte et de l'Enfant, CHU de Grenoble, Grenoble
  - Médecine - Consultations Douleur, CH de La Réole, La Réole
  - Unité Douleur et Soins Palliatifs, CH La Rochelle-Réaunis, La Rochelle
  - Pole enfant - CETD Salengro, CHRU de Lille, Lille
  - Pôle Anesthésie Consultation douleur, CHRU de Lille, Lille
  - CETD La Timone, AP-HM, Marseille
  - Centre d'Analgésie, CHRU Lapeyronie, Montpellier
  - Centre d'Evaluation et de Traitement de la Douleur, CHU de Nîmes, Nîmes
  - Service de Médecine de la Douleur et de Médecine Palliative, Hôpital Lariboisière-APHP, Paris
  - Service de lutte contre la douleur et d'Anesthésie, CH Périgueux, Périgueux
  - Service d'Explorations Fonctionnelles et Consultations Neurologiques, CH Lyon-Sud, Pierre-Bénite
  - Centre Antidouleurs, CHU de Reims, Reims
  - Centre de la Douleur, CHRU de Strasbourg, Strasbourg
  - Centre d'Analgésie Pédiatrique, Equipe Régionale Ressource en Soins Palliatifs-Equipe " Enfant-Do ", CHU de Toulouse, Toulouse
  - Centre d'évaluation et de traitement de la Douleur, Hôpital Pierre-Paul Ricquet, Toulouse

IPD SHARING:
Plan to Share IPD: No